CLINICAL TRIAL: NCT01945034
Title: Placebo-controlled, Double-blind Evaluation Of The Efficacy And Safety Of Ibuprofen 5% Topical Gel For The Treatment Of Ankle Sprain
Brief Title: 5% Topical Ibuprofen (IBU) for Ankle Sprain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B3491009
Record Dates: First submitted 2013-06-21; First posted 2013-09-18 (Estimated); Results first posted 2016-05-26 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-04

CONDITIONS: Ankle Injuries
Keywords: topical ibuprofen; ankle sprain
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Topical IBU twice daily (Experimental)
  Interventions: Drug: Topical IBU twice daily
- Placebo twice daily (Placebo Comparator)
  Interventions: Drug: Placebo twice daily
- Topical IBU three times daily (Experimental)
  Interventions: Drug: Topical IBU three times daily
- Placebo three times daily (Placebo Comparator)
  Interventions: Drug: Placebo three times daily

INTERVENTIONS:
Drug: Topical IBU twice daily — Topical gel administered as 4 inch strip twice daily for 7 days, and as needed for an additional 3 days
  Arms: Topical IBU twice daily
Drug: Placebo twice daily — Topical gel administered as a 4 inch strip twice daily for 7 days, and as needed for an additional 3 days
  Arms: Placebo twice daily
Drug: Topical IBU three times daily — Topical gel administered as a 4 inch strip three times daily for 7 days, and as needed for additional 3 days
  Arms: Topical IBU three times daily
Drug: Placebo three times daily — Topical gel administered as a 4 inch strip three times daily for 7 days, and as needed for additional 3 days
  Arms: Placebo three times daily

SUMMARY:
This study is being conducted to evaluate the effects of IBU 5% Topical Gel versus topical placebo for the relief of pain associated with a first or second degree ankle sprain. Both twice daily and three times daily regimens will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* First or second degree ankle sprain within 48 hours of first dose of study medication
* Medically cleared to participate

Exclusion Criteria:

* Similar injury of same joint within last 6 months
* Requires bed rest, surgery, or over-the-counter or prescription analgesics

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2013-11; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (19):
- United States (19):
  - Helen Keller Hospital, Sheffield, Alabama
  - Visions Clinical Research - Tucson, Tucson, Arizona
  - Orange County Research Institute, Anaheim, California
  - eStudy Site, San Diego, California
  - San Diego Sports Medicine and Family Health Center, San Diego, California
  - Sunrise Research Institute, Inc., Miami, Florida
  - L&L Research Choices, Miami, Florida
  - Doctors Research Network, South Miami, Florida
  - Elite Clinical Trials LLLP, Blackfoot, Idaho
  - MedPharmics, LLC, Metairie, Louisiana
  - Quality Clinical Research, Inc., Omaha, Nebraska
  - Heartland Clinical Research, Inc., Omaha, Nebraska
  - PMG Research of Salisbury, Salisbury, North Carolina
  - Lillestol Research, LLC, Fargo, North Dakota
  - Clinical Trial Network, Houston, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - Sports Medicine Associates of San Antonio, San Antonio, Texas
  - Danville Orthopedic Clinic, Danville, Virginia

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3491009&StudyName=5%25%20Topical%20Ibuprofen%20%28IBU%29%20for%20Ankle%20Sprain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted in United States from 08 November 2013 to 19 February 2015.
Pre-assignment Details: Out of the 348 screened participants, 304 were randomized and received treatment.
Groups:
- Ibuprofen Twice Daily: Ibuprofen 5 percent (%) topical gel twice daily was applied topically as a 4-inch strip approximately every 12 hours, for the first 7 days. Subsequently, on Days 8 through 10, participants were permitted to use the study medication on an optional basis, according to the assigned dosing regimen.
- Ibuprofen Thrice Daily: Ibuprofen 5% Topical Gel thrice a day was applied topically as a 4-inch strip approximately every 6 hours, for the first 7 days. Subsequently, on Days 8 through 10, participants were permitted to use the study medication on an optional basis, according to the assigned dosing regimen.
- Placebo Combined: Placebo matched to Ibuprofen twice daily or thrice daily regimen was applied for first 7 days.
Period: Overall Study
Arm/Group | Ibuprofen Twice Daily | Ibuprofen Thrice Daily | Placebo Combined
Started | 67 | 85 | 152
Completed | 66 | 80 | 145
Not Completed | 1 | 5 | 7
Not completed — Medication Error | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 1
Not completed — Other | 0 | 1 | 3
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Protocol Violation | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set included all randomized participants who dosed with the study medication and provided a baseline assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibuprofen Twice Daily | Ibuprofen Thrice Daily | Placebo Combined | Total
Number analyzed (Participants) | 67 | 85 | 152 | 304
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (15.20) | 35.2 (14.72) | 33.0 (13.90) | 33.3 (14.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 39 | 61 | 134
  Male | 33 | 46 | 91 | 170
Categorical Pain Severity Rating (PSR) [Number; unit: participants] — Participants were assessed by 4-Point category pain severity rating scale. Participants rated their pain upon weight bearing using a four-point scale, as follows: 0 = None, 1 = Mild, 2 = Moderate, 3 = Severe. All participants had moderate or severe ankle pain upon weight bearing at baseline.
  participants
    Moderate | 43 (1.25) | 63 (1.13) | 102 (1.17) | 208
    Severe | 24 | 22 | 50 | 96
Baseline Ankle Pain upon Weight Bearing [Mean (Standard Deviation); unit: Units on a scale] — Participants rated their pain on full weight-bearing movement. Pain Intensity (PI) was assessed on an 11-point numerical rating scale from 0=no pain to 10=most severe pain and this best describes their current pain in the injured ankle. At baseline, participants recorded a value of at least 6 (inclusive) to be eligible to participate in the study.
  Units on a scale | 8.3 (1.25) | 8.1 (1.13) | 8.4 (1.17) | 8.3 (1.18)
Baseline Ankle Pain at Rest [Mean (Standard Deviation); unit: Units on a scale] — Participants rated their pain at rest. PI was assessed on an 11-point numerical rating scale from 0=no pain to 10=most severe pain and this best describes their current pain in the injured ankle.
  Units on a scale | 6.2 (1.77) | 6.5 (1.48) | 6.5 (1.70) | 6.4 (1.65)
Baseline Participant's Global Assessment of Ankle Injury [Number; unit: participants] — Participants were asked the following question: "Considering all the ways your ankle injury affects you, how are you doing today?" The participant's response was recorded using a 5-point scale: 1 = Very Good, No symptoms and no limitations of normal activities; 2 = Good, Mild symptoms and no limitation of normal activities; 3 = Fair, Moderate symptoms and limitations of some normal activities; 4 = Poor, Severe symptoms and inability to carry out most normal activities; and 5 = Very Poor, Very severe symptoms which are intolerable and inability to carry out all normal activities.
  participants
    Very Good(1) | 0 | 0 | 0 | 0
    Good(2) | 0 | 0 | 7 | 7
    Fair(3) | 34 | 56 | 77 | 167
    Poor(4) | 30 | 25 | 55 | 110
    Very Poor(5) | 3 | 4 | 13 | 20
Baseline Physician Global Assessment of Ankle Injury [Number; unit: participants] — The physician assessment of the severity of the ankle injury was based on the participant's individual signs and symptoms which included pain, swelling, tenderness and limitation of range of movement, and graded using the following 6-point scale: 0 = Normal, No signs or symptoms; 1= Very mild, Very mild signs and symptoms; 2 = Mild, Mild signs and symptoms; 3 = Moderate, Moderate signs and symptoms; 4 = Severe, Severe signs and symptoms; 5 = Very severe, Very severe signs and symptoms.
  participants
    Normal(0) | 0 | 0 | 0 | 0
    Very mild(1) | 0 | 0 | 1 | 1
    Mild(2) | 9 | 28 | 30 | 67
    Moderate(3) | 50 | 54 | 101 | 205
    Severe(4) | 8 | 3 | 20 | 31
    Very severe(5) | 0 | 0 | 0 | 0
Baseline Participant Assessment of Normal Function/Activity [Number; unit: participants] — Participants were asked the following question: "How does your ankle injury affect your walking and normal activity?" The participant's response was recorded using a 5-point scale: 1=Normal activity and no pain; 2=Normal activity with pain; 3=Mildly restricted walking due to pain and can't resume normal activities; 4=Moderately restricted walking due to pain and can't resume normal activities; 5=Severely restricted walking due to pain and can't resume normal activities. The score ranges from 1-5, with higher scores indicates restricted activity.
  participants
    Normal walking/activity and no pain(1) | 0 | 0 | 0 | 0
    Normal walking/activity with pain(2) | 1 | 4 | 9 | 14
    Mild restrict walking(3) | 16 | 26 | 26 | 68
    Moderate restrict walking(4) | 43 | 45 | 91 | 179
    Severe restrict walking(5) | 7 | 10 | 26 | 43

OUTCOME MEASURES:

1. Primary Outcome: Sum of Pain Intensity Difference (SPID) on Weight Bearing Over 3 Days (SPID WB0-3)
Description: PI was assessed on an 11-point numerical rating scale from 0=no pain to 10=most severe pain. Pain intensity difference (PID) was the difference between baseline PI (prior to the first dose) and current PI at assessment. SPID was calculated as the time-weighted sum of PID scores over 3 days (72 hours). Total score ranges from -360 (higher pain relief) to 432 (lower pain relief) for SPID WB0-3. SPID is a value of change from baseline and as pain score at base line is usually higher than that at post baseline, a negative value of SPID indicates higher pain relief from baseline.
Time Frame: Over 3 Days (0-72 hours)
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ibuprofen Twice Daily | Ibuprofen Thrice Daily | Placebo Combined
Number analyzed (Participants) | 67 | 85 | 152
units on a scale | 188.9 (14.81) | 173.6 (13.6) | 165.9 (10.34)
Statistical Analysis 1: Comparison: Ibuprofen Twice Daily vs Placebo Combined; The analysis of variance (ANOVA) model was used which contains treatment, baseline categorical pain severity rating, pooled site blocks, and baseline pain intensity on weight bearing terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.190, ANOVA — p-value <=0.05 for treatment effects; LS Mean Difference = 23, 95% CI 2-sided [-11.49 to 57.56]
Statistical Analysis 2: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site blocks, and baseline pain intensity on weight bearing terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.633, ANOVA — p-value <=0.05 for treatment effects; LS Mean Difference = 7.8, 95% CI 2-sided [-24.20 to 39.70]
Statistical Analysis 3: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site blocks, and baseline pain intensity on weight bearing terms; Test type: Superiority or Other; p = 0.436, ANOVA — p-value <=0.05 for treatment effects; LS Mean Difference = -15.3, 95% CI 2-sided [-53.87 to 23.30]

2. Primary Outcome: Sum of Ankle Pain Intensity Difference on Weight Bearing Over 24 Hours After Dose 1 (SPID WB24)
Description: PI was assessed on an 11-point numerical rating scale from 0=no pain to 10=most severe pain. PID was the difference between baseline PI (prior to the first dose) and current PI at assessment. SPID was calculated as the time-weighted sum of PID scores over 24 hours. Total score ranges from -120 (higher pain relief) to 144 (lower pain relief) for SPID WB24. SPID is a value of change from baseline. Pain score at base line is usually higher than that at post baseline. So negative value of SPID indicates pain relief from baseline, while a positive value means a worst pain comparing to baseline, a negative value of SPID indicates higher pain relief from baseline.
Time Frame: 0 to 24 hours
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ibuprofen Twice Daily | Ibuprofen Thrice Daily | Placebo Combined
Number analyzed (Participants) | 67 | 85 | 152
units on a scale | 46.9 (5.03) | 41.1 (4.62) | 42.1 (3.51)
Statistical Analysis 1: Comparison: Ibuprofen Twice Daily vs Placebo Combined; The ANOVA model was used which contains treatment, baseline categorical pain severity rating (BLPSR), pooled site blocks, and baseline pain intensity on weight bearing (BLPIWB) terms. 95% CI not includes 0 for treatment effect. Upper limit of 95% CI< 0 for Ibuprofen treatment significantly better than combined Placebo. Comparison: tested at the 0.05 level of significance (2-sided). A comparison was eligible for being declared significant only if preceding comparison was significant; Test type: Superiority or Other; p = 0.426, ANOVA — p-value <=0.05 for treatment effects; Least Squares (LS) Mean Difference = 4.8, 95% CI 2-sided [-6.98 to 16.49]
Statistical Analysis 2: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; The ANOVA model was used which contains treatment, BLPSR, pooled site blocks, and BLPIWB terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo. Comparison: tested at the 0.05 level of significance (2-sided). A comparison was eligible for being declared significant only if preceding comparison was significant; Test type: Superiority or Other; p = 0.850, ANOVA — p-value <=0.05 for treatment effects; LS Mean Difference = -1.0, 95% CI 2-sided [-11.90 to 9.82]
Statistical Analysis 3: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; The ANOVA model was used which contains treatment, BLPSR, pooled site blocks, and BLPIWB terms. A comparison was eligible for being declared significant only if preceding comparison was significant; Test type: Superiority or Other; p = 0.385, ANOVA — p-value <=0.05 for treatment effects; LS Mean Difference = -5.8, 95% CI 2-sided [-18.91 to 7.32]

3. Secondary Outcome: Sum of Pain Intensity Difference at Rest Over 24 Hours on Day 1 (SPID R24)
Description: PI was assessed on an 11-point numerical rating scale from 0=no pain to 10=most severe pain. PID was the difference between baseline PI (prior to the first dose) and current PI at assessment. SPID was calculated as the time-weighted sum of PID scores over 24 hours. Total score ranges from -240 (higher pain relief) to 96 (lower pain relief) for SPID at rest. SPID is a value of change from baseline. Pain score at base line is usually higher than that at post baseline. So negative value of SPID indicates pain relief from baseline, while positive value means a worst pain comparing to baseline, a negative value of SPID indicates higher pain relief from baseline.
Time Frame: 0 to 24 hours
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ibuprofen Twice Daily | Ibuprofen Thrice Daily | Placebo Combined
Number analyzed (Participants) | 67 | 85 | 152
units on a scale | 44.7 (4.65) | 29.4 (4.29) | 34.7 (3.22)
Statistical Analysis 1: Comparison: Ibuprofen Twice Daily vs Placebo Combined; The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site blocks, and baseline pain intensity at rest terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.072, ANOVA — p-value <=0.05 for treatment effects; LS Mean Difference = 10, 95% CI 2-sided [-0.92 to 20.91]
Statistical Analysis 2: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.296, ANOVA — p-value <=0.05 for treatment effects; LS Mean Difference = -5.3, 95% CI 2-sided [-15.40 to 4.70]
Statistical Analysis 3: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site blocks, and baseline pain intensity at rest terms; Test type: Superiority or Other; p = 0.014, ANOVA — p-value <=0.05 for treatment effects; LS Mean Difference = -15.3, 95% CI 2-sided [-27.53 to -3.16]

4. Secondary Outcome: Change From Baseline in Participant's Global Assessment of Ankle Injury at Day 3 and 10
Description: Participant's global assessments of ankle injury was measured using 5-point scale: 1= Very Good (No symptoms and no limitations of normal activities), 2= Good (Mild symptoms and no limitation of normal activities), 3= Fair (Moderate symptoms and limitations of some normal activities), 4= Poor (Severe symptoms and inability to carry out most normal activities), 5= Very Poor (Very severe symptoms which are intolerable and inability to carry out all normal activities).
Time Frame: Baseline, Day 3, 10
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ibuprofen Twice Daily | Ibuprofen Thrice Daily | Placebo Combined
Number analyzed (Participants) | 67 | 85 | 152
units on a scale
  Change at: Day 3 | 0.7 (0.09) | 0.7 (0.08) | 0.6 (0.06)
  Change at: Day 10 | 1.8 (0.09) | 1.7 (0.09) | 1.6 (0.07)
Statistical Analysis 1: Comparison: Ibuprofen Twice Daily vs Placebo Combined; Day 3: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline participant global assessment terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.305, ANOVA — p-value <=0.05 for treatment effects; LS Mean Difference = 0.1, 95% CI 2-sided [-0.10 to 0.30]
Statistical Analysis 2: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.261, ANOVA — p-value <=0.05 for treatment effects; LS Mean Difference = 0.1, 95% CI 2-sided [-0.08 to 0.29]
Statistical Analysis 3: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; Day 3: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline participant global assessment terms; Test type: Superiority or Other; p = 0.996, ANOVA — p-value <=0.05 for treatment effects; LS Mean Difference = 0.0, 95% CI 2-sided [-0.22 to 0.22]
Statistical Analysis 4: Comparison: Ibuprofen Twice Daily vs Placebo Combined; Day 10: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline participant global assessment terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.210, ANOVA — p-value <=0.05 for treatment effects; LS Mean Difference = 0.1, 95% CI 2-sided [-0.08 to 0.36]
Statistical Analysis 5: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p = 0.556, ANOVA — p-value <=0.05 for treatment effects; LS Mean Difference = 0.1, 95% CI 2-sided [-0.14 to 0.27]
Statistical Analysis 6: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; Day 10: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline participant global assessment terms; Test type: Superiority or Other; p = 0.534, ANOVA — p-value <=0.05 for treatment effects; LS Mean Difference = -0.1, 95% CI 2-sided [-0.33 to 0.17]

5. Secondary Outcome: Change From Baseline in Physician Global Assessment of Ankle Injury at Day 3 and 10
Description: The physician assessment of the severity of the ankle injury was based on the participant's individual signs and symptoms which included pain, swelling, tenderness and limitation of range of movement, and was measured using 6-point scale: 0= Normal (No signs or symptoms) , 1= Very mild (Very mild signs and symptoms), 2= Mild (Mild signs and symptoms), 3= Moderate (Moderate signs and symptoms), 4= Severe (Severe signs and symptoms), 5= Very severe (Very severe signs and symptoms). A higher score is indicative of lesser improvement. Change from baseline was calculated as baseline value minus post-treatment value.
Time Frame: Baseline, Day 3, 10
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ibuprofen Twice Daily | Ibuprofen Thrice Daily | Placebo Combined
Number analyzed (Participants) | 67 | 85 | 152
units on a scale
  Change at: Day 3 | 0.7 (0.08) | 0.7 (0.07) | 0.8 (0.06)
  Change at: Day 10 | 1.8 (0.09) | 2.0 (0.09) | 2.0 (0.06)
Statistical Analysis 1: Comparison: Ibuprofen Twice Daily vs Placebo Combined; Day 3: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline physician global assessment terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.354, ANOVA — p-value <=0.05 for treatment effects; LS Mean Difference = -0.1, 95% CI 2-sided [-0.27 to 0.10]
Statistical Analysis 2: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; Day 3: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.237, ANOVA — p-value <=0.05 for treatment effects; LS Mean Difference = -0.1, 95% CI 2-sided [-0.28 to 0.07]
Statistical Analysis 3: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; Day 3: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline physician global assessment terms; Test type: Superiority or Other; p = 0.871, ANOVA — p-value <=0.05 for treatment effects; LS Mean Difference = -0.0, 95% CI 2-sided [-0.23 to 0.19]
Statistical Analysis 4: Comparison: Ibuprofen Twice Daily vs Placebo Combined; Day 10: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline physician global assessment terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.050, ANOVA — p-value <=0.05 for treatment effects; LS Mean Difference = -0.2, 95% CI 2-sided [-0.43 to -0.00]
Statistical Analysis 5: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 5, analysis 4]; Test type: Superiority or Other; p = 0.640, ANOVA — p-value <=0.05 for treatment effects; LS Mean Difference = -0.0, 95% CI 2-sided [-0.25 to 0.15]
Statistical Analysis 6: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; Day 10: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline physician global assessment terms; Test type: Superiority or Other; p = 0.180, ANOVA — p-value <=0.05 for treatment effects; LS Mean Difference = 0.2, 95% CI 2-sided [-0.08 to 0.41]

6. Secondary Outcome: Change From Baseline in Ankle Pain at Rest and Upon Weight Bearing (PID NRS) at Pre-specified Time Points
Description: PI in ankle pain at rest and upon weight bearing was assessed on an 11-point numerical rating scale from 0=no pain to 10=most severe pain. PID was the difference between baseline PI (prior to the first dose) and current PI at assessment. Pain score at baseline is usually higher than that at post baseline. So negative value of SPID indicates pain relief from baseline, while positive value means a worst pain comparing to baseline.
Time Frame: Baseline, 1, 2, 3, 4, 5, 6, 12(Day1),24(Day2),30(Day2),36(Day2),48(Day3),50(Day3),54(Day3),60(Day3),72(Day4),78(Day4),84(Day4), 96(Day5),102(Day5), 108 (Day5), 120(Day6),126(Day6),132(Day6),144(Day7),150(Day7),156(Day7) hours post first dose on Day 1
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ibuprofen Twice Daily | Ibuprofen Thrice Daily | Placebo Combined
Number analyzed (Participants) | 67 | 85 | 152
units on a scale
  Change at: At Rest 1 hour Day 1 | 1.3 (0.19) | 0.7 (0.17) | 1.2 (0.13)
  Change at: Upon Weight Bearing 1 hour Day 1 | 1.5 (0.20) | 1.1 (0.18) | 1.4 (0.14)
  Change at: At Rest 2 hour Day 1 | 1.7 (0.22) | 1.2 (0.20) | 1.5 (0.15)
  Change at: Upon Weight Bearing 2 hour Day 1 | 1.8 (0.23) | 1.5 (0.21) | 1.8 (0.16)
  Change at: At Rest 3 hour Day 1 | 1.9 (0.23) | 1.2 (0.22) | 1.6 (0.16)
  Change at: Upon Weight Bearing 3 hour Day 1 | 2.2 (0.25) | 1.7 (0.23) | 1.9 (0.17)
  Change at: At Rest 4 hour Day 1 | 1.8 (0.24) | 1.2 (0.22) | 1.5 (0.16)
  Change at: Upon Weight Bearing 4 hour Day 1 | 1.9 (0.25) | 1.8 (0.23) | 1.7 (0.18)
  Change at: At Rest 5 hour Day 1 | 1.9 (0.24) | 1.1 (0.22) | 1.4 (0.16)
  Upon Weight Bearing: 5 hour Day 1 | 2.2 (0.26) | 1.6 (0.24) | 1.7 (0.18)
  Change at: At Rest 6 hour Day 1 | 1.9 (0.24) | 1.1 (0.22) | 1.2 (0.16)
  Change at: Upon Weight Bearing 6 hour Day 1 | 2.1 (0.25) | 1.6 (0.23) | 1.5 (0.17)
  Change at: At Rest Day 1(PM) | 1.8 (0.22) | 1.1 (0.20) | 1.2 (0.15)
  Change at: Upon Weight Bearing Day 1(PM) | 2.0 (0.24) | 1.6 (0.22) | 1.6 (0.17)
  Change at: At Rest Day 2(AM) | 2.0 (0.22) | 1.3 (0.20) | 1.6 (0.15)
  Change at: Upon Weight Bearing Day 2(AM) | 2.0 (0.24) | 1.8 (0.22) | 1.9 (0.17)
  Change at: At Rest Day 2 Mid-day | 2.3 (0.23) | 1.7 (0.21) | 1.8 (0.16)
  Change at: Upon Weight Bearing Day 2 Mid-day | 2.5 (0.24) | 2.1 (0.22) | 2.1 (0.17)
  Change at: At Rest Day 2(PM) | 2.2 (0.23) | 1.9 (0.21) | 1.8 (0.16)
  Change at: Upon Weight Bearing Day 2(PM) | 2.4 (0.24) | 2.4 (0.22) | 2.1 (0.17)
  Change at: At Rest Day 3(AM) | 2.7 (0.22) | 2.0 (0.21) | 2.1 (0.16)
  Change at: Upon Weight Bearing Day 3(AM) | 2.8 (0.25) | 2.7 (0.23) | 2.5 (0.17)
  Change at: At Rest Day 3(AM + 2 hours) | 2.8 (0.24) | 2.2 (0.22) | 2.2 (0.16)
  Change at: Upon Weight Bearing Day 3(AM + 2 hours) | 2.9 (0.26) | 2.9 (0.24) | 2.6 (0.18)
  Change at: At Rest Day 3 Mid-day | 3.0 (0.23) | 2.2 (0.22) | 2.3 (0.16)
  Change at: Upon Weight Bearing Day 3 Mid-day | 3.2 (0.26) | 2.9 (0.24) | 2.7 (0.18)
  Change at: At Rest Day 3(PM) | 3.0 (0.23) | 2.1 (0.22) | 2.3 (0.16)
  Change at: Upon Weight Bearing Day 3(PM) | 3.1 (0.25) | 2.8 (0.23) | 2.7 (0.18)
  Change at: At Rest Day 4(AM) | 3.2 (0.23) | 2.5 (0.21) | 2.6 (0.16)
  Change at: Upon Weight Bearing Day 4(AM) | 3.4 (0.25) | 3.2 (0.23) | 3.0 (0.18)
  Change at: At Rest Day 4 Mid-day | 3.2 (0.25) | 2.5 (0.23) | 2.5 (0.17)
  Change at: Upon Weight Bearing Day 4 Mid-day | 3.5 (0.27) | 3.3 (0.25) | 3.2 (0.19)
  Change at: At Rest Day 4(PM) | 3.2 (0.24) | 2.7 (0.22) | 2.5 (0.17)
  Change at: Upon Weight Bearing Day 4(PM) | 3.4 (0.27) | 3.4 (0.25) | 3.1 (0.19)
  Change at: At Rest Day 5(AM) | 3.3 (0.24) | 2.8 (0.22) | 2.7 (0.17)
  Change at: Upon Weight Bearing Day 5(AM) | 3.7 (0.27) | 3.5 (0.24) | 3.3 (0.19)
  Change at: At Rest Day 5 Mid-day | 3.4 (0.25) | 2.9 (0.23) | 2.7 (0.17)
  Change at: Upon Weight Bearing Day 5 Mid-day | 3.7 (0.27) | 3.7 (0.25) | 3.3 (0.19)
  Change at: At Rest Day 5(PM) | 3.4 (0.25) | 3.0 (0.23) | 2.8 (0.17)
  Change at: Upon Weight Bearing Day 5(PM) | 3.8 (0.28) | 3.7 (0.26) | 3.5 (0.19)
  Change at: At Rest Day 6(AM) | 3.5 (0.25) | 3.2 (0.23) | 3.1 (0.17)
  Change at: Upon Weight Bearing Day 6(AM) | 3.9 (0.28) | 4.0 (0.26) | 3.8 (0.20)
  Change at: At Rest Day 6 Mid-day | 3.5 (0.25) | 3.3 (0.23) | 3.1 (0.17)
  Change at: Upon Weight Bearing Day 6 Mid-day | 3.8 (0.28) | 4.1 (0.26) | 3.7 (0.20)
  Change at: At Rest Day 6(PM) | 3.6 (0.26) | 3.3 (0.24) | 2.9 (0.18)
  Change at: Upon Weight Bearing Day 6(PM) | 3.9 (0.29) | 4.2 (0.27) | 3.7 (0.20)
  Change at: At Rest Day 7(AM) | 3.6 (0.25) | 3.5 (0.23) | 3.1 (0.17)
  Change at: Upon Weight Bearing Day 7(AM) | 4.2 (0.29) | 4.5 (0.27) | 3.9 (0.20)
  Change at: At Rest Day 7 Mid-day | 4.0 (0.25) | 3.6 (0.23) | 3.2 (0.18)
  Change at: Upon Weight Bearing Day 7 Mid-day | 4.6 (0.29) | 4.5 (0.27) | 4.1 (0.20)
  Change at: At Rest Day 7(PM) | 3.9 (0.25) | 3.7 (0.23) | 3.4 (0.17)
  Change at: Upon Weight Bearing Day 7(PM) | 4.5 (0.29) | 4.7 (0.27) | 4.2 (0.20)
Statistical Analysis 1: Comparison: Ibuprofen Twice Daily vs Placebo Combined; At Rest 1 hour Day 1: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.771, ANOVA; LS Mean Difference = 0.1, 95% CI 2-sided [-0.38 to 0.51]
Statistical Analysis 2: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.022, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.5, 95% CI 2-sided [-0.88 to -0.07]
Statistical Analysis 3: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; At Rest 1 hour Day 1: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms; Test type: Superiority or Other; p = 0.032, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.5, 95% CI 2-sided [-1.03 to -0.05]
Statistical Analysis 4: Comparison: Ibuprofen Twice Daily vs Placebo Combined; Upon Weight Bearing 1 hour Day 1: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.720, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.1, 95% CI 2-sided [-0.38 to 0.55]
Statistical Analysis 5: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p = 0.194, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.3, 95% CI 2-sided [-0.71 to 0.15]
Statistical Analysis 6: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; Upon Weight Bearing 1 hour Day 1: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms; Test type: Superiority or Other; p = 0.163, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.4, 95% CI 2-sided [-0.89 to 0.15]
Statistical Analysis 7: Comparison: Ibuprofen Twice Daily vs Placebo Combined; At Rest 2 hour Day 1: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.644, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.1, 95% CI 2-sided [-0.40 to 0.64]
Statistical Analysis 8: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p = 0.129, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.4, 95% CI 2-sided [-0.85 to 0.11]
Statistical Analysis 9: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; At Rest 2 hour Day 1: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms; Test type: Superiority or Other; p = 0.096, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.5, 95% CI 2-sided [-1.07 to 0.09]
Statistical Analysis 10: Comparison: Ibuprofen Twice Daily vs Placebo Combined; Upon Weight Bearing 2 hour Day 1: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.905, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.0, 95% CI 2-sided [-0.50 to 0.57]
Statistical Analysis 11: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.279, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.3, 95% CI 2-sided [-0.77 to 0.22]
Statistical Analysis 12: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; Upon Weight Bearing 2 hour Day 1: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms; Test type: Superiority or Other; p = 0.315, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.3, 95% CI 2-sided [-0.90 to 0.29]
Statistical Analysis 13: Comparison: Ibuprofen Twice Daily vs Placebo Combined; At Rest 3 hour Day 1: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.203, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.4, 95% CI 2-sided [-0.19 to 0.91]
Statistical Analysis 14: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 13]; Test type: Superiority or Other; p = 0.207, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.3, 95% CI 2-sided [-0.83 to 0.18]
Statistical Analysis 15: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; At Rest 3 hour Day 1: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms; Test type: Superiority or Other; p = 0.030, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.7, 95% CI 2-sided [-1.30 to -0.07]
Statistical Analysis 16: Comparison: Ibuprofen Twice Daily vs Placebo Combined; Upon Weight Bearing 3 hour Day 1: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.372, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.3, 95% CI 2-sided [-0.32 to 0.84]
Statistical Analysis 17: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 16]; Test type: Superiority or Other; p = 0.532, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.2, 95% CI 2-sided [-0.70 to 0.36]
Statistical Analysis 18: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; Upon Weight Bearing 3 hour Day 1: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms; Test type: Superiority or Other; p = 0.189, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.4, 95% CI 2-sided [-1.08 to 0.21]
Statistical Analysis 19: Comparison: Ibuprofen Twice Daily vs Placebo Combined; At Rest 4 hour Day 1: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.264, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.3, 95% CI 2-sided [-0.24 to 0.87]
Statistical Analysis 20: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; At Rest 4 hour Day 1:The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.260, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.3, 95% CI 2-sided [-0.81 to 0.22]
Statistical Analysis 21: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; At Rest 4 hour Day 1: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms; Test type: Superiority or Other; p = 0.054, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.6, 95% CI 2-sided [-1.23 to 0.01]
Statistical Analysis 22: Comparison: Ibuprofen Twice Daily vs Placebo Combined; Upon Weight Bearing 4 hour Day 1: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.456, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.2, 95% CI 2-sided [-0.37 to 0.81]
Statistical Analysis 23: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 22]; Test type: Superiority or Other; p = 0.639, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.1, 95% CI 2-sided [-0.42 to 0.68]
Statistical Analysis 24: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; Upon Weight Bearing 4 hour Day 1: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms; Test type: Superiority or Other; p = 0.780, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.1, 95% CI 2-sided [-0.75 to 0.57]
Statistical Analysis 25: Comparison: Ibuprofen Twice Daily vs Placebo Combined; At Rest 5 hour Day 1: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.071, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.5, 95% CI 2-sided [-0.04 to 1.07]
Statistical Analysis 26: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 25]; Test type: Superiority or Other; p = 0.468, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.2, 95% CI 2-sided [-0.70 to 0.32]
Statistical Analysis 27: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; At Rest 5 hour Day 1: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms; Test type: Superiority or Other; p = 0.027, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.7, 95% CI 2-sided [-1.33 to -0.08]
Statistical Analysis 28: Comparison: Ibuprofen Twice Daily vs Placebo Combined; Upon Weight Bearing 5 hour Day 1: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.107, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.5, 95% CI 2-sided [-0.11 to 1.09]
Statistical Analysis 29: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 28]; Test type: Superiority or Other; p = 0.947, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.0, 95% CI 2-sided [-0.57 to 0.53]
Statistical Analysis 30: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; Upon Weight Bearing 5 hour Day 1: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms; Test type: Superiority or Other; p = 0.134, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.5, 95% CI 2-sided [-1.18 to 0.16]
Statistical Analysis 31: Comparison: Ibuprofen Twice Daily vs Placebo Combined; At Rest 6 hour Day 1: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.017, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.7, 95% CI 2-sided [0.12 to 1.23]
Statistical Analysis 32: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 31]; Test type: Superiority or Other; p = 0.715, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.1, 95% CI 2-sided [-0.60 to 0.41]
Statistical Analysis 33: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; At Rest 6 hour Day 1: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms; Test type: Superiority or Other; p = 0.015, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.8, 95% CI 2-sided [-1.39 to -0.15]
Statistical Analysis 34: Comparison: Ibuprofen Twice Daily vs Placebo Combined; Upon Weight Bearing 6 hour Day 1: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.027, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.7, 95% CI 2-sided [0.07 to 1.23]
Statistical Analysis 35: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 34]; Test type: Superiority or Other; p = 0.660, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.1, 95% CI 2-sided [-0.42 to 0.65]
Statistical Analysis 36: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; Upon Weight Bearing 6 hour Day 1: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms; Test type: Superiority or Other; p = 0.107, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.5, 95% CI 2-sided [-1.18 to 0.11]
Statistical Analysis 37: Comparison: Ibuprofen Twice Daily vs Placebo Combined; At Rest Day 1(PM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.020, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.6, 95% CI 2-sided [0.10 to 1.13]
Statistical Analysis 38: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 37]; Test type: Superiority or Other; p = 0.749, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.1, 95% CI 2-sided [-0.55 to 0.40]
Statistical Analysis 39: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; At Rest Day 1(PM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms; Test type: Superiority or Other; p = 0.019, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.7, 95% CI 2-sided [-1.27 to -0.12]
Statistical Analysis 40: Comparison: Ibuprofen Twice Daily vs Placebo Combined; Upon Weight Bearing Day 1(PM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.163, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.4, 95% CI 2-sided [-0.16 to 0.96]
Statistical Analysis 41: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 40]; Test type: Superiority or Other; p = 0.727, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.1, 95% CI 2-sided [-0.43 to 0.61]
Statistical Analysis 42: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; Upon Weight Bearing Day 1(PM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms; Test type: Superiority or Other; p = 0.336, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.3, 95% CI 2-sided [-0.94 to 0.32]
Statistical Analysis 43: Comparison: Ibuprofen Twice Daily vs Placebo Combined; At Rest Day 2(AM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.174, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.4, 95% CI 2-sided [-0.16 to 0.87]
Statistical Analysis 44: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 43]; Test type: Superiority or Other; p = 0.277, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.3, 95% CI 2-sided [-0.73 to 0.21]
Statistical Analysis 45: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; At Rest Day 2(AM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms; Test type: Superiority or Other; p = 0.035, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.6, 95% CI 2-sided [-1.19 to -0.04]
Statistical Analysis 46: Comparison: Ibuprofen Twice Daily vs Placebo Combined; Upon Weight Bearing Day 2(AM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.858, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.1, 95% CI 2-sided [-0.50 to 0.60]
Statistical Analysis 47: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 46]; Test type: Superiority or Other; p = 0.724, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.1, 95% CI 2-sided [-0.60 to 0.42]
Statistical Analysis 48: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; Upon Weight Bearing Day 2(AM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms; Test type: Superiority or Other; p = 0.651, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.1, 95% CI 2-sided [-0.76 to 0.48]
Statistical Analysis 49: Comparison: Ibuprofen Twice Daily vs Placebo Combined; At Rest Day 2 Mid-day: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.059, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.5, 95% CI 2-sided [-0.02 to 1.05]
Statistical Analysis 50: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 49]; Test type: Superiority or Other; p = 0.766, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.1, 95% CI 2-sided [-0.57 to 0.42]
Statistical Analysis 51: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; At Rest Day 2 Mid-day: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms; Test type: Superiority or Other; p = 0.053, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.6, 95% CI 2-sided [-1.19 to 0.01]
Statistical Analysis 52: Comparison: Ibuprofen Twice Daily vs Placebo Combined; Upon Weight Bearing Day 2 Mid-day: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.212, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.4, 95% CI 2-sided [-0.21 to 0.92]
Statistical Analysis 53: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 52]; Test type: Superiority or Other; p = 0.911, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.0, 95% CI 2-sided [-0.49 to 0.55]
Statistical Analysis 54: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; Upon Weight Bearing Day 2 Mid-day: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms; Test type: Superiority or Other; p = 0.305, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.3, 95% CI 2-sided [-0.96 to 0.30]
Statistical Analysis 55: Comparison: Ibuprofen Twice Daily vs Placebo Combined; At Rest Day 2(PM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.075, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.5, 95% CI 2-sided [-0.05 to 1.02]
Statistical Analysis 56: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 55]; Test type: Superiority or Other; p = 0.684, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.1, 95% CI 2-sided [-0.39 to 0.60]
Statistical Analysis 57: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; At Rest Day 2(PM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms; Test type: Superiority or Other; p = 0.208, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.4, 95% CI 2-sided [-0.98 to 0.21]
Statistical Analysis 58: Comparison: Ibuprofen Twice Daily vs Placebo Combined; Upon Weight Bearing Day 2(PM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.304, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.3, 95% CI 2-sided [-0.27 to 0.85]
Statistical Analysis 59: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 58]; Test type: Superiority or Other; p = 0.356, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.2, 95% CI 2-sided [-0.27 to 0.76]
Statistical Analysis 60: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; Upon Weight Bearing Day 2(PM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms; Test type: Superiority or Other; p = 0.876, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.0, 95% CI 2-sided [-0.67 to 0.58]
Statistical Analysis 61: Comparison: Ibuprofen Twice Daily vs Placebo Combined; At Rest Day 3(AM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.020, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.6, 95% CI 2-sided [0.10 to 1.15]
Statistical Analysis 62: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 61]; Test type: Superiority or Other; p = 0.940, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.0, 95% CI 2-sided [-0.50 to 0.47]
Statistical Analysis 63: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; At Rest Day 3(AM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms; Test type: Superiority or Other; p = 0.032, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.6, 95% CI 2-sided [-1.23 to -0.06]
Statistical Analysis 64: Comparison: Ibuprofen Twice Daily vs Placebo Combined; Upon Weight Bearing Day 3(AM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.206, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.4, 95% CI 2-sided [-0.21 to 0.95]
Statistical Analysis 65: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; Upon Weight Bearing Day 3(AM):The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.310, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.3, 95% CI 2-sided [-0.26 to 0.81]
Statistical Analysis 66: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; Upon Weight Bearing Day 3(AM):The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms; Test type: Superiority or Other; p = 0.771, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.1, 95% CI 2-sided [-0.74 to 0.55]
Statistical Analysis 67: Comparison: Ibuprofen Twice Daily vs Placebo Combined; At Rest Day 3(AM + 2 hours): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.016, ANOVA; p-value <=0.05 for treatment effects; LS Mean difference = 0.7, 95% CI 2-sided [0.13 to 1.24]
Statistical Analysis 68: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 67]; Test type: Superiority or Other; p = 0.905, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.0, 95% CI 2-sided [-0.48 to 0.54]
Statistical Analysis 69: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; At Rest Day 3(AM + 2 hours): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms; Test type: Superiority or Other; p = 0.039, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.7, 95% CI 2-sided [-1.28 to -0.03]
Statistical Analysis 70: Comparison: Ibuprofen Twice Daily vs Placebo Combined; Upon Weight Bearing Day 3(AM + 2 hours): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.276, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.3, 95% CI 2-sided [-0.27 to 0.93]
Statistical Analysis 71: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 70]; Test type: Superiority or Other; p = 0.343, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.3, 95% CI 2-sided [-0.29 to 0.82]
Statistical Analysis 72: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; Upon Weight Bearing Day 3(AM + 2 hours): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms; Test type: Superiority or Other; p = 0.849, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.1, 95% CI 2-sided [-0.73 to 0.60]
Statistical Analysis 73: Comparison: Ibuprofen Twice Daily vs Placebo Combined; At Rest Day 3 Mid-day: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.009, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.7, 95% CI 2-sided [0.19 to 1.29]
Statistical Analysis 74: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 73]; Test type: Superiority or Other; p = 0.763, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.1, 95% CI 2-sided [-0.58 to 0.43]
Statistical Analysis 75: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; At Rest Day 3 Mid-day: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms; Test type: Superiority or Other; p = 0.010, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.8, 95% CI 2-sided [-1.43 to -0.20]
Statistical Analysis 76: Comparison: Ibuprofen Twice Daily vs Placebo Combined; Upon Weight Bearing Day 3 Mid-day: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.105, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.5, 95% CI 2-sided [-0.10 to 1.09]
Statistical Analysis 77: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 76]; Test type: Superiority or Other; p = 0.533, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.2, 95% CI 2-sided [-0.38 to 0.73]
Statistical Analysis 78: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; Upon Weight Bearing Day 3 Mid-day: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms; Test type: Superiority or Other; p = 0.348, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.3, 95% CI 2-sided [-0.99 to 0.35]
Statistical Analysis 79: Comparison: Ibuprofen Twice Daily vs Placebo Combined; At Rest Day 3(PM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.016, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.7, 95% CI 2-sided [0.13 to 1.23]
Statistical Analysis 80: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 79]; Test type: Superiority or Other; p = 0.483, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.2, 95% CI 2-sided [-0.69 to 0.33]
Statistical Analysis 81: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; At Rest Day 3(PM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms; Test type: Superiority or Other; p = 0.006, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.9, 95% CI 2-sided [-1.47 to -0.25]
Statistical Analysis 82: Comparison: Ibuprofen Twice Daily vs Placebo Combined; Upon Weight Bearing Day 3(PM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.177, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.4, 95% CI 2-sided [-0.19 to 1.00]
Statistical Analysis 83: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 82]; Test type: Superiority or Other; p = 0.586, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.2, 95% CI 2-sided [-0.40 to 0.70]
Statistical Analysis 84: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; Upon Weight Bearing Day 3(PM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms; Test type: Superiority or Other; p = 0.448, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.3, 95% CI 2-sided [-0.92 to 0.41]
Statistical Analysis 85: Comparison: Ibuprofen Twice Daily vs Placebo Combined; At Rest Day 4(AM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.043, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.6, 95% CI 2-sided [0.02 to 1.09]
Statistical Analysis 86: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 85]; Test type: Superiority or Other; p = 0.688, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.1, 95% CI 2-sided [-0.59 to 0.39]
Statistical Analysis 87: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; At Rest Day 4(AM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms; Test type: Superiority or Other; p = 0.032, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.7, 95% CI 2-sided [-1.25 to -0.06]
Statistical Analysis 88: Comparison: Ibuprofen Twice Daily vs Placebo Combined; Upon Weight Bearing Day 4(AM):The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.179, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.4, 95% CI 2-sided [-0.19 to 0.99]
Statistical Analysis 89: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; Upon Weight Bearing Day 4(AM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.609, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.1, 95% CI 2-sided [-0.40 to 0.69]
Statistical Analysis 90: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; Upon Weight Bearing Day 4(AM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms; Test type: Superiority or Other; p = 0.435, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.3, 95% CI 2-sided [-0.92 to 0.40]
Statistical Analysis 91: Comparison: Ibuprofen Twice Daily vs Placebo Combined; At Rest Day 4 Mid-day: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.023, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.7, 95% CI 2-sided [0.10 to 1.26]
Statistical Analysis 92: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 91]; Test type: Superiority or Other; p = 0.987, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.0, 95% CI 2-sided [-0.54 to 0.53]
Statistical Analysis 93: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; At Rest Day 4 Mid-day: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms; Test type: Superiority or Other; p = 0.040, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.7, 95% CI 2-sided [-1.33 to -0.03]
Statistical Analysis 94: Comparison: Ibuprofen Twice Daily vs Placebo Combined; Upon Weight Bearing Day 4 Mid-day: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.319, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.3, 95% CI 2-sided [-0.31 to 0.94]
Statistical Analysis 95: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 94]; Test type: Superiority or Other; p = 0.712, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.1, 95% CI 2-sided [-0.47 to 0.69]
Statistical Analysis 96: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; Upon Weight Bearing Day 4 Mid-day: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms; Test type: Superiority or Other; p = 0.557, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.2, 95% CI 2-sided [-0.91 to 0.49]
Statistical Analysis 97: Comparison: Ibuprofen Twice Daily vs Placebo Combined; At Rest Day 4(PM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.015, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.7, 95% CI 2-sided [0.14 to 1.28]
Statistical Analysis 98: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 97]; Test type: Superiority or Other; p = 0.326, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.3, 95% CI 2-sided [-0.26 to 0.79]
Statistical Analysis 99: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; At Rest Day 4(PM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms; Test type: Superiority or Other; p = 0.167, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.4, 95% CI 2-sided [-1.08 to 0.19]
Statistical Analysis 100: Comparison: Ibuprofen Twice Daily vs Placebo Combined; Upon Weight Bearing Day 4(PM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.350, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.3, 95% CI 2-sided [-0.33 to 0.93]
Statistical Analysis 101: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 100]; Test type: Superiority or Other; p = 0.235, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.4, 95% CI 2-sided [-0.23 to 0.93]
Statistical Analysis 102: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; Upon Weight Bearing Day 4(PM):The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms; Test type: Superiority or Other; p = 0.881, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.1, 95% CI 2-sided [-0.65 to 0.76]
Statistical Analysis 103: Comparison: Ibuprofen Twice Daily vs Placebo Combined; At Rest Day 5(AM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.036, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.6, 95% CI 2-sided [0.04 to 1.16]
Statistical Analysis 104: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 103]; Test type: Superiority or Other; p = 0.656, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.1, 95% CI 2-sided [-0.40 to 0.63]
Statistical Analysis 105: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; At Rest Day 5(AM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms; Test type: Superiority or Other; p = 0.130, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.5, 95% CI 2-sided [-1.11 to 0.14]
Statistical Analysis 106: Comparison: Ibuprofen Twice Daily vs Placebo Combined; Upon Weight Bearing Day 5(AM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.304, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.3, 95% CI 2-sided [-0.30 to 0.95]
Statistical Analysis 107: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; Upon Weight Bearing Day 5(AM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms; Test type: Superiority or Other; p = 0.491, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.2, 95% CI 2-sided [-0.37 to 0.78]
Statistical Analysis 108: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; [analysis description as in outcome 6, analysis 107]; Test type: Superiority or Other; p = 0.726, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.1, 95% CI 2-sided [-0.82 to 0.57]
Statistical Analysis 109: Comparison: Ibuprofen Twice Daily vs Placebo Combined; At Rest Day 5 Mid-day: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.029, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.6, 95% CI 2-sided [0.07 to 1.23]
Statistical Analysis 110: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 109]; Test type: Superiority or Other; p = 0.585, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.1, 95% CI 2-sided [-0.39 to 0.68]
Statistical Analysis 111: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; At Rest Day 5 Mid-day: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms; Test type: Superiority or Other; p = 0.131, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.5, 95% CI 2-sided [-1.15 to 0.15]
Statistical Analysis 112: Comparison: Ibuprofen Twice Daily vs Placebo Combined; Upon Weight Bearing Day 5 Mid-day: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.215, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.4, 95% CI 2-sided [-0.24 to 1.04]
Statistical Analysis 113: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 112]; Test type: Superiority or Other; p = 0.244, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.3, 95% CI 2-sided [-0.24 to 0.94]
Statistical Analysis 114: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; Upon Weight Bearing Day 5 Mid-day: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms; Test type: Superiority or Other; p = 0.885, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.1, 95% CI 2-sided [-0.76 to 0.66]
Statistical Analysis 115: Comparison: Ibuprofen Twice Daily vs Placebo Combined; At Rest Day 5(PM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.067, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.5, 95% CI 2-sided [-0.04 to 1.13]
Statistical Analysis 116: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 115]; Test type: Superiority or Other; p = 0.500, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.2, 95% CI 2-sided [-0.35 to 0.73]
Statistical Analysis 117: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; At Rest Day 5(PM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms; Test type: Superiority or Other; p = 0.276, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.4, 95% CI 2-sided [-1.02 to 0.29]
Statistical Analysis 118: Comparison: Ibuprofen Twice Daily vs Placebo Combined; Upon Weight Bearing Day 5(PM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.413, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.3, 95% CI 2-sided [-0.38 to 0.92]
Statistical Analysis 119: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 118]; Test type: Superiority or Other; p = 0.448, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.2, 95% CI 2-sided [-0.37 to 0.83]
Statistical Analysis 120: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; Upon Weight Bearing Day 5(PM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms; Test type: Superiority or Other; p = 0.917, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.0, 95% CI 2-sided [-0.76 to 0.69]
Statistical Analysis 121: Comparison: Ibuprofen Twice Daily vs Placebo Combined; At Rest Day 6(AM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.132, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.4, 95% CI 2-sided [-0.13 to 1.03]
Statistical Analysis 122: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 121]; Test type: Superiority or Other; p = 0.505, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.2, 95% CI 2-sided [-0.35 to 0.72]
Statistical Analysis 123: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; At Rest Day 6(AM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms; Test type: Superiority or Other; p = 0.422, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.3, 95% CI 2-sided [-0.92 to 0.38]
Statistical Analysis 124: Comparison: Ibuprofen Twice Daily vs Placebo Combined; Upon Weight Bearing Day 6(AM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.747, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.1, 95% CI 2-sided [-0.54 to 0.76]
Statistical Analysis 125: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 124]; Test type: Superiority or Other; p = 0.386, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.3, 95% CI 2-sided [-0.34 to 0.87]
Statistical Analysis 126: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; Upon Weight Bearing Day 6(AM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms; Test type: Superiority or Other; p = 0.668, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.2, 95% CI 2-sided [-0.57 to 0.89]
Statistical Analysis 127: Comparison: Ibuprofen Twice Daily vs Placebo Combined; At Rest Day 6 Mid-day: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.099, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.5, 95% CI 2-sided [-0.09 to 1.08]
Statistical Analysis 128: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 127]; Test type: Superiority or Other; p = 0.365, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.2, 95% CI 2-sided [-0.29 to 0.79]
Statistical Analysis 129: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; At Rest Day 6 Mid-day: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms; Test type: Superiority or Other; p = 0.463, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.2, 95% CI 2-sided [-0.90 to 0.41]
Statistical Analysis 130: Comparison: Ibuprofen Twice Daily vs Placebo Combined; Upon Weight Bearing Day 6 Mid-day: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.845, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.1, 95% CI 2-sided [-0.60 to 0.73]
Statistical Analysis 131: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 130]; Test type: Superiority or Other; p = 0.199, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.4, 95% CI 2-sided [-0.21 to 1.02]
Statistical Analysis 132: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; Upon Weight Bearing Day 6 Mid-day: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms; Test type: Superiority or Other; p = 0.375, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.3, 95% CI 2-sided [-0.41 to 1.08]
Statistical Analysis 133: Comparison: Ibuprofen Twice Daily vs Placebo Combined; At Rest Day 6(PM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.028, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.7, 95% CI 2-sided [0.07 to 1.27]
Statistical Analysis 134: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 133]; Test type: Superiority or Other; p = 0.188, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.4, 95% CI 2-sided [-0.18 to 0.92]
Statistical Analysis 135: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; At Rest Day 6(PM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms; Test type: Superiority or Other; p = 0.375, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.3, 95% CI 2-sided [-0.97 to 0.37]
Statistical Analysis 136: Comparison: Ibuprofen Twice Daily vs Placebo Combined; Upon Weight Bearing Day 6(PM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.552, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.2, 95% CI 2-sided [-0.47 to 0.89]
Statistical Analysis 137: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 136]; Test type: Superiority or Other; p = 0.126, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.5, 95% CI 2-sided [-0.14 to 1.12]
Statistical Analysis 138: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; Upon Weight Bearing Day 6(PM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms; Test type: Superiority or Other; p = 0.460, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.3, 95% CI 2-sided [-0.47 to 1.05]
Statistical Analysis 139: Comparison: Ibuprofen Twice Daily vs Placebo Combined; At Rest Day 7(AM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.095, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.5, 95% CI 2-sided [-0.09 to 1.09]
Statistical Analysis 140: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 139]; Test type: Superiority or Other; p = 0.146, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.4, 95% CI 2-sided [-0.14 to 0.94]
Statistical Analysis 141: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; At Rest Day 7(AM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms; Test type: Superiority or Other; p = 0.769, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.1, 95% CI 2-sided [-0.75 to 0.56]
Statistical Analysis 142: Comparison: Ibuprofen Twice Daily vs Placebo Combined; Upon Weight Bearing Day 7(AM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.405, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.3, 95% CI 2-sided [-0.39 to 0.96]
Statistical Analysis 143: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 142]; Test type: Superiority or Other; p = 0.073, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.6, 95% CI 2-sided [-0.05 to 1.20]
Statistical Analysis 144: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; Upon Weight Bearing Day 7(AM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms; Test type: Superiority or Other; p = 0.458, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.3, 95% CI 2-sided [-0.47 to 1.04]
Statistical Analysis 145: Comparison: Ibuprofen Twice Daily vs Placebo Combined; At Rest Day 7 Mid-day: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.009, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.8, 95% CI 2-sided [0.20 to 1.39]
Statistical Analysis 146: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 145]; Test type: Superiority or Other; p = 0.209, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.4, 95% CI 2-sided [-0.20 to 0.90]
Statistical Analysis 147: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; At Rest Day 7 Mid-day: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms; Test type: Superiority or Other; p = 0.193, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.4, 95% CI 2-sided [-1.11 to 0.22]
Statistical Analysis 148: Comparison: Ibuprofen Twice Daily vs Placebo Combined; Upon Weight Bearing Day 7 Mid-day: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.149, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.5, 95% CI 2-sided [-0.18 to 1.18]
Statistical Analysis 149: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 148]; Test type: Superiority or Other; p = 0.186, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.4, 95% CI 2-sided [-0.21 to 1.06]
Statistical Analysis 150: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; Upon Weight Bearing Day 7 Mid-day: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms; Test type: Superiority or Other; p = 0.845, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.1, 95% CI 2-sided [-0.84 to 0.69]
Statistical Analysis 151: Comparison: Ibuprofen Twice Daily vs Placebo Combined; At Rest Day 7(PM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.067, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.5, 95% CI 2-sided [-0.04 to 1.14]
Statistical Analysis 152: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 151]; Test type: Superiority or Other; p = 0.242, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.3, 95% CI 2-sided [-0.22 to 0.87]
Statistical Analysis 153: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; At Rest Day 7(PM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms; Test type: Superiority or Other; p = 0.498, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.2, 95% CI 2-sided [-0.88 to 0.43]
Statistical Analysis 154: Comparison: Ibuprofen Twice Daily vs Placebo Combined; Upon Weight Bearing Day 7(PM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.330, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.3, 95% CI 2-sided [-0.34 to 1.02]
Statistical Analysis 155: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 6, analysis 154]; Test type: Superiority or Other; p = 0.124, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.5, 95% CI 2-sided [-0.14 to 1.13]
Statistical Analysis 156: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; Upon Weight Bearing Day 7(PM): The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms; Test type: Superiority or Other; p = 0.687, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.2, 95% CI 2-sided [-0.61 to 0.92]

7. Secondary Outcome: Sum of Pain Intensity Difference at Rest and on Weight Bearing Over 6 Hours on Day 1 and Over 2 Hours on Day 3
Description: PI at rest and on weight bearing was assessed on an 11-point numerical rating scale from 0=no pain to 10=most severe pain. PID was the difference between baseline PI (prior to the first dose) and current PI at assessment. SPID 0-6 was calculated as the time-weighted sum of PID scores over 6 hours on Day 1, with a total score ranges from -30 (higher pain relief) to 36 (lower pain relief). SPID 0-12 was calculated as the time weighted sum of PID scores over 2 hours on Day 3, with a total score ranges from -10 (higher pain relief) to 12 (lower pain relief). SPID is a value of change from baseline. Pain score at base line is usually higher than that at post baseline. So negative value of SPID indicates pain relief from baseline, while positive value means a worst pain comparing to baseline, a negative value of SPID indicates higher pain relief from baseline.
Time Frame: Over 6 hours on Day 1, over 2 hours on Day 3
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ibuprofen Twice Daily | Ibuprofen Thrice Daily | Placebo Combined
Number analyzed (Participants) | 67 | 85 | 152
units on a scale
  At Rest over 6 Hours on Day 1 | 10.4 (1.24) | 6.6 (1.14) | 8.4 (0.86)
  Weight Bearing over 6 Hours on Day 1 | 11.7 (1.31) | 9.4 (1.20) | 9.9 (0.91)
  At Rest over 2 Hours on Day 3 | 109.6 (9.54) | 79.4 (8.80) | 84.7 (6.60)
  Weight Bearing over 2 Hours on Day 3 | 116.1 (10.11) | 106.8 (9.29) | 102.4 (7.06)
Statistical Analysis 1: Comparison: Ibuprofen Twice Daily vs Placebo Combined; At Rest over 6 Hours on Day 1: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.166, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 2.0, 95% CI 2-sided [-0.85 to 4.95]
Statistical Analysis 2: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.199, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -1.7, 95% CI 2-sided [-4.42 to 0.93]
Statistical Analysis 3: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; At Rest over 6 Hours on Day 1: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms; Test type: Superiority or Other; p = 0.022, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -3.8, 95% CI 2-sided [-7.04 to -0.56]
Statistical Analysis 4: Comparison: Ibuprofen Twice Daily vs Placebo Combined; Weight Bearing over 6 Hours on Day 1: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.260, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 1.7, 95% CI 2-sided [-1.30 to 4.79]
Statistical Analysis 5: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 7, analysis 4]; Test type: Superiority or Other; p = 0.729, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.5, 95% CI 2-sided [-3.31 to 2.32]
Statistical Analysis 6: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; Weight Bearing over 6 Hours on Day 1: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms; Test type: Superiority or Other; p = 0.196, ANOVA; LS Mean Difference = -2.2, 95% CI 2-sided [-5.64 to 1.16]
Statistical Analysis 7: Comparison: Ibuprofen Twice Daily vs Placebo Combined; At Rest over 2 Hours on Day 3: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.030, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 24.9, 95% CI 2-sided [2.49 to 47.28]
Statistical Analysis 8: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; p = 0.018, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -30.2, 95% CI 2-sided [-55.24 to -5.23]
Statistical Analysis 9: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; At Rest over 2 Hours on Day 3: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms; Test type: Superiority or Other; p = 0.611, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -5.3, 95% CI 2-sided [-25.98 to 15.29]
Statistical Analysis 10: Comparison: Ibuprofen Twice Daily vs Placebo Combined; Weight Bearing over 2 Hours on Day 3: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.251, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 13.8, 95% CI 2-sided [-9.80 to 37.36]
Statistical Analysis 11: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 7, analysis 10]; Test type: Superiority or Other; p = 0.689, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 4.4, 95% CI 2-sided [-17.37 to 26.26]
Statistical Analysis 12: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; Weight Bearing over 2 Hours on Day 3: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms; Test type: Superiority or Other; p = 0.486, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -9.3, 95% CI 2-sided [-35.69 to 17.01]

8. Secondary Outcome: Sum of Pain Intensity Difference Scores at Rest Over 3 Days
Description: PI was assessed on an 11-point numerical rating scale from 0=no pain to 10=most severe pain. PID was the difference between baseline PI (prior to the first dose) and current PI at assessment. SPID was calculated as the time-weighted sum of PID scores over 3 days (72 hours). Total score ranges from -360 (higher pain relief) to 432 (lower pain relief). SPID is a value of change from baseline. Pain score at base line is usually higher than that at post baseline. So negative value of SPID indicates pain relief from baseline, while positive value means a worst pain comparing to baseline, a negative value of SPID indicates higher pain relief from baseline.
Time Frame: Over 3 Days (0-72 hours)
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Ibuprofen Twice Daily | Ibuprofen Thrice Daily | Placebo Combined
Number analyzed (Participants) | 67 | 85 | 152
Units on a scale | 177.6 (13.90) | 131.1 (12.83) | 139.0 (9.62)
Statistical Analysis 1: Comparison: Ibuprofen Twice Daily vs Placebo Combined; At Rest Over 3 Days: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.021, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 38.5, 95% CI 2-sided [5.90 to 71.18]
Statistical Analysis 2: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.603, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -7.9, 95% CI 2-sided [-38.02 to 22.12]
Statistical Analysis 3: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; At Rest Over 3 Days: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms; Test type: Superiority or Other; p = 0.013, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -46.5, 95% CI 2-sided [-82.93 to -10.05]

9. Secondary Outcome: Sum of Pain Intensity Difference Scores at Rest and on Weight Bearing Over 7 Days
Description: PI was assessed on an 11-point numerical rating scale from 0=no pain to 10=most severe pain. PID was the difference between baseline PI (prior to the first dose) and current PI at assessment. SPID was calculated as the time-weighted sum of PID scores over 7 days (168 hours). Total score ranges from -840 (higher pain relief) to 1008 (lower pain relief). SPID is a value of change from baseline. Pain score at baseline is usually higher than that at post baseline. So negative value of SPID indicates pain relief from baseline, while positive value means a worst pain comparing to baseline, a negative value of SPID indicates higher pain relief from baseline.
Time Frame: Over 7 days (0-168 hours)
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Ibuprofen Twice Daily | Ibuprofen Thrice Daily | Placebo Combined
Number analyzed (Participants) | 67 | 85 | 152
Units on a scale
  At Rest: Over 7 Days | 472.5 (31.60) | 396.6 (29.16) | 384.8 (21.88)
  Weight Bearing: Over 7 Days | 516.4 (34.52) | 507.7 (31.70) | 470.4 (24.09)
Statistical Analysis 1: Comparison: Ibuprofen Twice Daily vs Placebo Combined; At Rest Over 7 days: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.021, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 87.7, 95% CI 2-sided [13.48 to 161.85]
Statistical Analysis 2: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.735, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 11.8, 95% CI 2-sided [-56.59 to 80.11]
Statistical Analysis 3: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; At Rest Over 7 days: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity at rest terms; Test type: Superiority or Other; p = 0.072, ANOVA; LS Mean Difference = -75.9, 95% CI 2-sided [-158.73 to 6.93]
Statistical Analysis 4: Comparison: Ibuprofen Twice Daily vs Placebo Combined; Weight Bearing Over 7 Days: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.261, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 46.0, 95% CI 2-sided [-34.43 to 126.52]
Statistical Analysis 5: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 9, analysis 4]; Test type: Superiority or Other; p = 0.325, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 37.3, 95% CI 2-sided [-37.13 to 111.80]
Statistical Analysis 6: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; Weight Bearing Over 7 Days: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline pain intensity on weight bearing terms; Test type: Superiority or Other; p = 0.849, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -8.7, 95% CI 2-sided [-98.64 to 81.22]

10. Secondary Outcome: Change From Baseline in Participant Assessment of Normal Function and Activity at Day 3 and 10
Description: Participant assessment of normal function was measured using a 5-point scale: 1= Normal walking/activity and no pain; 2= Normal walking/activity with pain; 3= Mildly restricted walking due to pain and can't resume normal activities; 4= Moderately restricted walking due to pain and can't resume normal activities; 5= Severely restricted walking due to pain and can't resume normal activities. The normal functioning and activity scores for each question range from 1 to 5, with higher scores indicating worsening of normal activity.
Time Frame: Baseline, Day 3, 10
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Ibuprofen Twice Daily | Ibuprofen Thrice Daily | Placebo Combined
Number analyzed (Participants) | 67 | 85 | 152
Units on a scale
  Change at: Day 3 | 1.0 (0.10) | 0.9 (0.09) | 0.7 (0.07)
  Change at: Day 10 | 2.1 (0.07) | 2.1 (0.09) | 2.1 (0.09)
Statistical Analysis 1: Comparison: Ibuprofen Twice Daily vs Placebo Combined; Day 3: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline participant assessment of Normal Function/Activity terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.042, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.2, 95% CI 2-sided [0.0 to 0.49]
Statistical Analysis 2: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.114, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.2, 95% CI 2-sided [-0.04 to 0.40]
Statistical Analysis 3: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; Day 3: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline participant assessment of Normal Function/Activity terms; Test type: Superiority or Other; p = 0.598, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.1, 95% CI 2-sided [-0.34 to 0.20]
Statistical Analysis 4: Comparison: Ibuprofen Twice Daily vs Placebo Combined; Day 10: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline participant assessment of Normal Function/Activity terms. Upper limit of 95% CI < 0 for Ibuprofen treatment significantly better than combined Placebo; Test type: Superiority or Other; p = 0.833, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = -0.0, 95% CI 2-sided [-0.24 to 0.19]
Statistical Analysis 5: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 10, analysis 4]; Test type: Superiority or Other; p = 0.853, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.0, 95% CI 2-sided [-0.18 to 0.22]
Statistical Analysis 6: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; Day 10: The ANOVA model was used which contains treatment, baseline categorical pain severity rating, pooled site block, and baseline participant assessment of Normal Function/Activity terms; Test type: Superiority or Other; p = 0.733, ANOVA; p-value <=0.05 for treatment effects; LS Mean Difference = 0.0, 95% CI 2-sided [-0.20 to 0.29]

11. Secondary Outcome: Participant's Global Assessment of Medication at End of Study
Description: Participants Global Assessment of Medication was used to rate the medication as a pain reliever. The responses of participants were recorded using 5-point scale: 1= Very Poor, 2= Poor, 3= Fair, 4= Good, 5= Very Good. The global assessment of medication scores for each question range from 0 to 5, giving a possible score range of 0 - 5, with higher scores indicating medication as a better pain reliever.
Time Frame: Day 10
Population: The full analysis set included all randomized participants who dosed with the study medication and provided a baseline assessment. Number of participants analyzed 'N' signifies those participants who were evaluable for the measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ibuprofen Twice Daily | Ibuprofen Thrice Daily | Placebo Combined
Number analyzed (Participants) | 62 | 75 | 141
Units on a scale | 3.8 (1.18) | 4 (0.94) | 4 (1.03)

12. Secondary Outcome: Time to First Perceptible Relief and Meaningful Relief
Description: Participants evaluated time to first perceptible relief by stopping a stopwatch labelled 'first perceptible relief' at moment participant first began to experience any relief, exact question asked was: "Stop stopwatch when you first begin to feel any pain-relieving effect whatsoever of product; that is, when you first feel a little relief". First perceptible relief was considered confirmed by meaningful relief if participant achieved both "first perceptible" and "meaningful" relief by either pressing second stopwatch or by indicating that his/her "first perceptible" relief was also "meaningful". For "time to meaningful relief," exact question asked was: "Stop this stopwatch when you have meaningful relief; that is, when relief from pain is meaningful to you." Stopwatches were active up to 3 hours after dosing or until stopped by participant, or rescue medication was administered.
Time Frame: 0 to 3 hours on Day 1
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Ibuprofen Twice Daily | Ibuprofen Thrice Daily | Placebo Combined
Number analyzed (Participants) | 67 | 85 | 152
Minutes
  First Perceptible Relief | 12.9 [10.1 to 15.7] | 36.4 [24.7 to 56.4] | 22.7 [15.7 to 30.3]
  Meaningful Relief | 41.6 [31.6 to 67.5] | NA [NA to NA] — Median and Confidence interval (CI) was not analyzed, as median was greater than 180 minutes. | 72.6 [58.1 to 116.1]
Statistical Analysis 1: Comparison: Ibuprofen Twice Daily vs Placebo Combined; Time to First Perceptible Relief: Hazard Ratio and corresponding 95% CI were calculated based on the Wald statistic from the Proportional Hazards (PH) model with treatment, BLPSR, and pooled site blocks; Test type: Superiority or Other; p = 0.016, Proportional Hazards Model; p-value <=0.05 for treatment effects; Hazard Ratio (HR) = 1.45, 95% CI 2-sided [1.07 to 1.97]
Statistical Analysis 2: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; Time to First Perceptible Relief: Hazard Ratio and corresponding 95% CI were calculated based on the Wald statistic from the PH model with treatment, BLPSR, and pooled site blocks; Test type: Superiority or Other; p = 0.022, Proportional Hazards Model; p-value <=0.05 for treatment effects; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.53 to 0.95]
Statistical Analysis 3: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; [analysis description as in outcome 12, analysis 2]; Test type: Superiority or Other; p < 0.001, Proportional Hazards Model; p-value <=0.05 for treatment effects; Hazard Ratio (HR) = 0.49, 95% CI 2-sided [0.34 to 0.69]
Statistical Analysis 4: Comparison: Ibuprofen Twice Daily vs Placebo Combined; Time to Meaningful Relief: Hazard Ratio and corresponding 95% CI were calculated based on the Wald statistic from the PH model with treatment, BLPSR, and pooled site blocks; Test type: Superiority or Other; p < 0.001, Proportional Hazards Model; p-value <=0.05 for treatment effects; Hazard Ratio (HR) = 1.79, 95% CI 2-sided [1.27 to 2.51]
Statistical Analysis 5: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; [analysis description as in outcome 12, analysis 4]; Test type: Superiority or Other; p = 0.009, Proportional Hazards Model; p-value <=0.05 for treatment effects; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.41 to 0.88]
Statistical Analysis 6: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; [analysis description as in outcome 12, analysis 4]; Test type: Superiority or Other; p < 0.001, Proportional Hazards Model; p-value <=0.05 for treatment effects; Hazard Ratio (HR) = 0.34, 95% CI 2-sided [0.22 to 0.52]

13. Secondary Outcome: Time to Rescue Medication After Initial Dose, and After Each Subsequent Dose
Description: Participants used only acetaminophen at a dose of 500 milligram (mg) every 6 hours product as needed (PRN) as rescue medication during the course of the study. Participants who used acetaminophen were to record its use, and date and time of administration in the participant diary. Time to rescue medication after initial dose, after each subsequent dose, provided that in each dose interval at least 25% of the participants take rescue medication was analyzed using the proportional hazard model with site, treatment group, and baseline categorical ankle pain terms in the model.
Time Frame: Post-Dose on Day 1 up to Day 10
Population: Data was not analyzed since <20% participants used rescue medication.
Arm/Group | Ibuprofen Twice Daily | Ibuprofen Thrice Daily | Placebo Combined
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Number of Doses of Rescue Medication Used During the First 7 Days of Dosing
Description: Participants received only acetaminophen 500 mg every 6 hours PRN as rescue medication during the course of the study.
Time Frame: Baseline up to Day 7
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Doses
Arm/Group | Ibuprofen Twice Daily | Ibuprofen Thrice Daily | Placebo Combined
Number analyzed (Participants) | 67 | 85 | 152
Doses | 1.7 (3.83) | 0.6 (1.41) | 1.2 (3.96)
Statistical Analysis 1: Comparison: Ibuprofen Twice Daily vs Placebo Combined; Test type: Superiority or Other; p = 0.479, Cochran-Mantel-Haenszel; p-values from the Cochran-Mantel-Haenszel (CMH) test with modified ridit scores, controlling for BLPSR and site block
Statistical Analysis 2: Comparison: Ibuprofen Thrice Daily vs Placebo Combined; Test type: Superiority or Other; p = 0.279, Cochran-Mantel-Haenszel; p-values from the CMH test with modified ridit scores, controlling for BLPSR and site block
Statistical Analysis 3: Comparison: Ibuprofen Twice Daily vs Ibuprofen Thrice Daily; Test type: Superiority or Other; p = 0.129, Cochran-Mantel-Haenszel; p-values from the CMH test with modified ridit scores, controlling for BLPSR and site block

15. Secondary Outcome: Percentage of Participants Taking Rescue Medication
Description: Participants used only acetaminophen at a dose of 500 mg every 6 hours PRN as analgesia or rescue therapy during the course of the study. Participants who used acetaminophen were to record its use, and date and time of administration in the participant diary.
Time Frame: Post first dose Day 1 up to Day 10
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Ibuprofen Twice Daily | Ibuprofen Thrice Daily | Placebo Combined
Number analyzed (Participants) | 67 | 85 | 152
Percentage of participants | 28.4 | 18.8 | 25.7

ADVERSE EVENTS:
Time Frame: Baseline up to 14 days after last study drug dose administration (Day 10)
Arm/Group | Ibuprofen Twice Daily | Ibuprofen Thrice Daily | Placebo Combined
Serious Adverse Events (participants affected / at risk) | 1/67 | 0/85 | 0/152
Other Adverse Events (participants affected / at risk) | 4/67 | 5/85 | 13/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ibuprofen Twice Daily (N=67) | Ibuprofen Thrice Daily (N=85) | Placebo Combined (N=152)
Pregnancy of partner (Social circumstances) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ibuprofen Twice Daily (N=67) | Ibuprofen Thrice Daily (N=85) | Placebo Combined (N=152)
Eye irritation (Eye disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 1 | 0 | 1
Application site erythema (General disorders) | 0 | 0 | 1
Influenza like illness (General disorders) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 4
Dizziness (Nervous system disorders) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Sticky skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.